CLINICAL TRIAL: NCT02991586
Title: Effectiveness Study of a Dialectical Behavioral Treatment for Adolescents With Emotional Instability and Their Families. Comparison of Family Functioning and Cope Strategies in Adolescents With Emotional Instability and Their Families and a Control Group
Brief Title: Effectiveness Study of a Dialectical Behavioral Treatment for Adolescents With Emotional Instability and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, María Mayoral, Clinical Psychologist, Hospital General Universitario Gregorio Marañon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FALGregorioMaranon
Record Dates: First submitted 2016-06-10; First posted 2016-12-13 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Emotional Instability
Keywords: Emotional Instability; Family Therapy; BPD; DBT
MeSH Terms: interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialectical Behavior Therapy (Experimental): Dialectical Behavior Therapy (DBT) is a cognitive behavioral treatment that was originally developed to treat chronically suicidal individuals diagnosed with borderline personality disorder (BPD) and it is now recognized as the gold standard psychological treatment for this population. In addition, research has shown that it is effective in treating a wide range of other disorders such as substance dependence, depression, post-traumatic stress disorder (PTSD), and eating disorders. In this research DBT skills will be taught to parents of adolescents with high emotional instability
  Interventions: Behavioral: Dialectical Behaviour Therapy
- Control (No Intervention): Control: The "No intervention arm" in this research is defined as follow:, sons and daughters are in their respective treatment but parents are nor receiving any DBT intervention

INTERVENTIONS:
Behavioral: Dialectical Behaviour Therapy — Group of families
  Arms: Dialectical Behavior Therapy

SUMMARY:
Emotional instability disorder (IE) is appreciable since adolescence, and crises (suicidal ideation, self-harm, impulsive acts and brief psychotic episodes) carry a high use of health resources, coupled with the suffering of families who feel helpless and difficulties in handling.

this study is composed of three diferents studies:

. The first study's goal is to determine if there are diferences and, which ones, between family functioning and cope strategies between adolescents with IE and their families, and families of a control group.

* the purpose of the second study is to evaluate the effectivenes of a dialectical behavior therapy for adolescents with IE and their families who are in treatment in the Child Abd Adolescent Mental Heath Service of the Hospital sant Joan de Déu Terres de Lleida. This treatment consist on 2 preliminary sessions with parents and patients and 12 group sessions which purpose is to teach skilss to manage emotions based on dialectical Behavior Therapy.
* finally, the third study is designed to evaluate the effectiveness of a dialectical behavior therapy (DBT) for parents of adolescents with IE who are in treatment in the different network devices of Child and Adolescent Mental Health of the Community of Madrid. Treatment goals are the development of communication skills, validation and crisis management as well as increase understanding and competence of the pathology. The DBT intervention will begin with two individual sessions with parents of patients and 10 theoretical and practical seminars in group format (6-7 families) following the model proposed by Marsha Linehan. The DBT interventions will be added to "standard treatment" that a patient with IE receives in the investigative devices.

DETAILED DESCRIPTION:
* In the first study, case group is composed by patients with IE and their families, both from Madrid and Lérida. The control group is composed by adolescents without mental pathologies, recruited from some high scholls from Madrid and Lérida.
* In the second study, the results will be measured a after the end of treatment and 6 months after the treatment ends.

In the third study, the results will be measured a after the end of treatment and 6 months after the treatment ends.

ELIGIBILITY:
Inclusion Criteria:

* Parents of patients aged 12-17 years whose child is at least 3 criteria of borderline personality disorder ( Diagnostic and Statistical Manual of Mental Disorders 5 ) .
* Talk correctly Spanish correctly.
* Coexistence with son and willingness to participate in the groups.
* Informed consent.

Exclusion Criteria:

* Mental retardation.
* Being involved in some other structured DBT family intervention.
* Parents whose children are not receiving any treatment .
* Participated in Actions for Treatment of Personality in Adolescence (ATRAPA TAI)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2016-05; Primary Completion 2022-01 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotional Regulation Scale (DERS). (Hervás 2008) | one year
Automatic Anger and Hostility Thoughts Scale (IPRI) (Magán 2010) | one year
Coping Styles and Strategies Scale (COPE) (Crespo 1997) | one year

SECONDARY OUTCOMES:
Children Relapses and Self harms Questionnaire (Ad Hoc) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mayoral, PhD, Principal Investigator — Gregorio Marañon Hospital
Locations (1):
- Instituto Provincial de Psiquiatria, Hospital General Universitario Gregorio Maranon. Calle Ibiza 43, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793